CLINICAL TRIAL: NCT05852756
Title: The Effect of Nutrition Education Given by Pecha Kucha Method on Preventing Malnutrition to Cancer Patients Receiving Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Gülcan Bahçecioğlu Turan, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/ 03- 23
Record Dates: First submitted 2023-05-01; First posted 2023-05-10 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Preventing Malnutrition

STUDY DESIGN:
Intervention Model Description: pecha kucha training
Who Masked: Participant
Masking Description: Single (Participant) preventing malnutrition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: (Experimental): pecha kucha will be practiced
  Interventions: Behavioral: pecha kucha
- control (No Intervention): Routine maintenance will be applied.

INTERVENTIONS:
Behavioral: pecha kucha — pecha kucha training
  Arms: Experimental:

SUMMARY:
The leading goal of cancer treatment is to eradicate the cancer. If the primary goal is not achieved, it is aimed to prolong life, improve quality of life, or improve symptoms. Cancer treatments are divided into two basic groups as local and systemic. Systemic treatments include chemotherapy, hormone therapy, targeted molecular therapy, immunotherapy treatments. Local treatments are; ablative approaches that include surgery, cryotherapy, radiotherapy and radiofrequency. Radiotherapy (RT) is a treatment method in which ionizing beam is used. The aim of radiotherapy in cancer treatment is to destroy the tumor, if this is not possible, to provide palliative treatment. Radiotherapy uses ionizing radiation in the form of electromagnetic waves (x-rays, gamma rays) or particles for this purpose. Pecha Kucha (PK), meaning "chat voice" or "chat" in Japanese, refers to a well-crafted, fast and concise presentation format. In a PK presentation, each presenter is only allowed to show 20 PowerPoint slides for 20 seconds each on a timer. In other words, the presenter has only 20 seconds to discuss each slide before the next slide appears, and the presentation time is limited to 6 minutes and 40 seconds. Ideas are explained visually with pictures and graphics, and slides have little text.

DETAILED DESCRIPTION:
According to the report of the World Health Organization, the increase in cancer is predicted to be over 70% by 2020 in developing countries.

While a significant increase in the life span of cancer patients has been achieved with effective multi-faceted treatment approaches in recent years, nutritional problems related to cancer and cancer treatment have begun to emerge as an important factor in quality of life and survival. Early detection of nutritional disorders and initiation of necessary nutritional support are of great importance in increasing the effect of radiotherapy and chemotherapy, reducing infection rates, increasing clinical response and life expectancy. Pecha Kucha (PK), meaning "chat voice" or "chat" in Japanese, refers to a well-crafted, fast and concise presentation format. In a PK presentation, each presenter is only allowed to show 20 PowerPoint slides for 20 seconds each on a timer. In other words, the presenter has only 20 seconds to discuss each slide before the next slide appears, and the presentation time is limited to 6 minutes and 40 seconds. Ideas are explained visually with pictures and graphics, and slides have little text.

ELIGIBILITY:
Inclusion Criteria:

* • Patients over 18 years of age

  * Patients receiving radiotherapy for the first time
  * Patients with cachectic and diagnosed mental problems
  * Patients who can read and write or who can get support from their relatives
  * Patients who can be contacted

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
NRS-2002 (Nutritional Risk Screening) Evaluation Form | 1 hours later
  The development of scale was done with a different method compared to the development of other scanning tools. The scoring system consists of two parts as 'nutritional status' and 'disease severity' and provides scoring as 'no problem', 'mild', 'moderate' and 'severe'. Scoring is made between 0-3 for each section. In addition to scoring in patients over the age of seventy, 1 more point is added to the score due to age. Patients with a total score of ≥3 are considered to be at nutritional risk.
Subjective Global Assessment (SGD) | 1 hours later
  The Subjectif Global Assessment scale (SGD) is a clinical technique that is described based on anamnesis and physical examination characteristics. The major components of SGD are weight loss in the last 6 months and weight loss in the last 2 weeks. In the physical examination, it is questioned whether there is loss of subcutaneous adipose tissue, muscle wasting, ankle/scrotal edema and ascites. The history is taken from the patient, if possible, or from a family member if not. It is very important to consider the primary disease and the nutritional requirements associated with the disease. The clinician should be unaware of the patient's laboratory findings in terms of the subjective nature of the method in SGD.
  After recording the parameters related to the subjective global assessment, the patient is evaluated in three categories: 'well-nourished' (A), 'moderately or suspected malnourished' (B) and 'severely malnourished' (C).

CONTACTS AND LOCATIONS:
Locations (1):
- Gülcan B.Turan, Elâzığ, Merkez, Turkey (Türkiye)

REFERENCES:
- [Derived] Bahcecioglu Turan G, Karaaslan F, Ozer Z. The effects of nutrition education with Pecha Kucha method on prevention of malnutrition in cancer patients undergoing radiotherapy: a randomised controlled study. BMC Cancer. 2025 Aug 22;25(1):1355. doi: 10.1186/s12885-025-14626-7. PMID 40847291